CLINICAL TRIAL: NCT02070068
Title: A Pilot Study to Optimize Imaging When Utilizing the PINPOINT Endoscopic Fluorescence Imaging System for Identification of Biliary Anatomy During Laparoscopic Biliary and Hepatic Operations
Brief Title: A Pilot Dosing and Timing Study to Optimize Imaging When Utilizing Endoscopic Fluorescence Imaging System During Laparoscopic Biliary and Hepatic Operations
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Principal Investigator, Ali Zarrinpar, Assistant Professor, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PP LBH 01
Record Dates: First submitted 2014-02-19; First posted 2014-02-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Biliary Anatomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): ICG administered 10 minutes prior to time of visualization
  Interventions: Device: PINPOINT System
- Group 2 (Experimental): ICG administered 45 min prior to time of visualization
  Interventions: Device: PINPOINT System

INTERVENTIONS:
Device: PINPOINT System

SUMMARY:
Operations on the liver, bile ducts, and gallbladders are some of the most commonly performed abdominal operations in the United States. Cholecystectomy, removal of the gallbladder, is the most common of these with more than 750,000 performed annually. Injury to the common bile duct (CBD) during these procedures occur infrequently (approximately 0.1% to 0.5%), but it is an important source of patient morbidity. Serious injuries often require at least one surgical repair, and these repairs have variable long-term outcomes. Techniques to allow the visualization of the bile ducts may prevent such an injury, by providing vital information about the presence of gallstones in the CBD and show a surgical road map of the ducts. Near-infrared (NIR) cholangiography has the advantage over standard cholangiography of not exposing patients and healthcare providers to radiation. This technique also allows the superimposition of the cholangiogram onto the normal image.

This study is being conducted to optimize an imaging technique called PINPOINT. Images will be obtained during clinically necessary operations. The images will be evaluated to determine the best method for locating and outlining the anatomy. The information learned will guide the future use of PINPOINT in laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, subjects must fulfill all of the following criteria:

1. Subjects who are healthy men or women 18 years of age or older.
2. Subjects who are scheduled for laparoscopic biliary or hepatic operations.
3. Subjects who sign an approved informed consent form for the study.
4. Subjects who are willing to comply with the protocol.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subjects with a known allergy or history of adverse reaction to ICG, iodine or iodine dyes.
2. Subjects who, in the Investigator's opinion, have any medical condition that makes the subject a poor candidate for the investigational procedure, or interferes with the interpretation of study results.
3. Subjects who are pregnant or lactating females.
4. Subjects, who are actively participating in another investigational clinical study and who, in the Investigator's or Sponsor's opinion, should not be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Ease of Identification of Biliary Anatomy as Scored by the Surgeon (1-5 scale) | 10 minutes after injection
Ease of Identification of Biliary Anatomy as Scored by the Surgeon (1-5 scale) | 45 minutes after injection

CONTACTS AND LOCATIONS:
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States